CLINICAL TRIAL: NCT03967847
Title: Oral Ketorolac as an Adjuvant Agent for Postoperative Pain Control Following Arthroscopic Rotator Cuff Repair
Brief Title: Oral Ketorolac for Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Robert J. Gillespie, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180949
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Rotator Cuff Tear; Postoperative Pain
Keywords: Rotator Cuff Tear; Postoperative Pain
MeSH Terms: conditions — Rotator Cuff Injuries; Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (No Intervention)
- Ketorolac (Experimental)
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Oral Ketorolac
  Arms: Ketorolac

SUMMARY:
1. The investigators aim to examine the use of IV and oral ketorolac as an adjunctive agent to the standard of care pain protocol for postoperative pain control following arthroscopic rotator cuff repair.
2. The investigators hypothesize that the use of IV and oral ketorolac in addition to the standard of care pain protocol will reduce postoperative opioid consumption following arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria

1. Patients between the ages of 18 and 89 years old, male or female
2. Patients undergoing primary shoulder arthroscopic rotator cuff repair

Exclusion Criteria

1. Patients below the age of 18 or above the age of 89
2. Illiterate or non-English speaking patients
3. Patients with contraindications to Ketorolac
4. History of alcohol of drug abuse
5. Chronic use of analgesic or psychotropic drugs
6. Known peptic ulcer disease or bleeding diathesis
7. Renal dysfunction

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 patients were enrolled/randomized but only 39 patients were included for final analysis because of incomplete data collection
Groups:
- Control: Control: no ketorolac
Period: Overall Study
Arm/Group | Control | Ketorolac
Started | 21 | 23
Completed | 21 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 44 patients were enrolled/randomized but only 39 patients were included for final analysis because of incomplete data collection
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (12.9) | 55.7 (8.2) | 55.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 11 | 15 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 15 | 27
  Black | 7 | 5 | 12
  Hispanic | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Other | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (6.1) | 32.9 (6.5) | 31 (6.3)
Smoker [Count of Participants; unit: Participants] | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Visual Analog Scale Scores
Description: The Visual Analog Scale ranges from a minimum score of 0 to a maximum score of 100. A smaller score would be considered a better outcome.
Time Frame: participants were assessed at one single time point up to 8 weeks.
Measure: Median (Inter-Quartile Range); unit: score/units on a scale
Groups:
- Control: No ketorolac
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 19 | 20
score/units on a scale | 30 [15 to 50] | 20 [8.75 to 32.5]

2. Secondary Outcome: Number of Participants With Retear of Rotator Cuff Repair
Description: Assessing retear of rotator cuff repair on postop MRI.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 11 | 11
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 14 months
Description: The time frame that is expressed is that over which each participant was assessed
Arm/Group | Control | Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 16/19 | 9/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=19) | Ketorolac (N=20)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) — Nausea/Vomiting
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Drowsiness (Nervous system disorders) | 4 (4) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Itching (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT03967847/Prot_SAP_000.pdf